CLINICAL TRIAL: NCT05429879
Title: The Impact of Music on Pain and Anxiety During Flexible Cystoscopies: A Comparison Between the Patient's Preferred Music, Classical Music, and the Absence of Music
Brief Title: The Impact of Music on Pain and Anxiety During Flexible Cystoscopies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Horizon Health Network (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Gavin Langille, Staff Urologist, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101548
Record Dates: First submitted 2022-05-26; First posted 2022-06-23 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Flexible Cystoscopy
Keywords: Flexible cystoscopy; Music therapy; Urology; Anxiety; Pain; Satisfaction; Discomfort; Preferred music; Classical music
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized control study that is designed to study outcomes between subjects. Participants will be randomly assigned to one of three groups and will be stratified according to sex. Stratified randomization will be done by selection of sequential pre-filled envelopes containing the group for a particular patient at the time of cystoscopy - This is a 1:1:1 randomization with equal group membership performed for both male and female sexes - The envelopes will be randomized by pre-assigning an order of participants to each of the three groups within each sex using a Random sequence generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preferred Music Arm (Experimental): This arm will allow patients to listen to their preferred music choice during their cystoscopy.
  Interventions: Other: Preferred Music Arm
- Classical Music Arm (Experimental): Patients will listen to a standard playlist of copyright free classical music.
  Interventions: Other: Classical Music Arm
- No music Arm (No Intervention): Patients will not listen to music during cystoscopy.

INTERVENTIONS:
Other: Preferred Music Arm — Patients will choose their preferred music to be played during the cystoscopy procedure. No music will be played prior to or immediately after the flexible cystoscopy procedure. Music will be delivered via a speaker allowing for communication between the urologist and the patient during the procedure. Aside from addition of music, standard of care will not be impacted.
  Arms: Preferred Music Arm
Other: Classical Music Arm — A standardized playlist of copyright free classical music will be played during the cystoscopy procedure. No music will be played prior to or immediately after the flexible cystoscopy procedure. Music will be delivered via a speaker allowing for communication between the urologist and the patient during the procedure. Aside from addition of music, standard of care will not be impacted.
  Arms: Classical Music Arm

SUMMARY:
Background: Cystoscopy is a routine diagnostic test often performed in the outpatient Urology setting. However, patients may sometimes feel pain and anxiety during this procedure. Distraction therapies, including patient preferred music and classical music may reduce pain and anxiety associated with cystoscopy. However, it is unclear if patient preferred music has greater positive outcomes for patients than classical music.

Hypothesis: We hypothesize that patient preferred music during flexible cystoscopies will reduce patient self-reported pain and anxiety scores when compared to classical music and absence of music.

Objective: To assess whether a patient's preferred music reduces pain and anxiety during cystoscopies when compared to classical music and the absence of music Methods: This is a prospective randomized control study where patients undergoing flexible cystoscopy in the outpatient Urology clinic will be randomly assigned to one of three groups: Preferred music, classical music, or no music for their procedure. Differences in pain and anxiety will be assessed between groups using the Visual Analog Scale and State-Trait Anxiety Inventory scale.

Potential Benefits: Identifying and understanding non-pharmacological interventions that can reduce pain and anxiety during cystoscopies is an important task that will allow urologists to better manage these patients.

DETAILED DESCRIPTION:
Previous studies have shown that using music as a non-pharmacological intervention is an effective, safe, and inexpensive way to address pain and anxiety in patients during cystoscopies. However few studies have compared patient outcomes between preferred music and classical music groups, and no studies have compared these groups in a North American sample population. The intent of this project is to compare pain and anxiety in those listening to their preferred music, classical music, and no music during their cystoscopy to assess what might be the optimal way to provide this non-pharmacological intervention. Identifying and understanding non-pharmacological interventions that can reduce pain and anxiety during cystoscopies is an important task that will allow urologists to better manage these patients. The purpose of this study is to assess the impact of a patient's preferred choice of music on pain and anxiety when compared to classical music and the absence of music.

The study design will included a 1:1:1 randomization with equal group membership performed for both male and female sexes. Group 1 will allow patients to listen to their preferred music choice during cystoscopy, group 2 will listen to a standardized copyright free playlist of classical music, and group 3 will listen to no music and serve as a control group. Patients will be recruited and consented on the day of the procedure prior to filling out the State Trait Anxiety Inventory (STAI) questionnaire. After their procedure, patients will fill out the STAI questionnaire; Visual Analog Scales (VAS) for pain, satisfaction, and discomfort; and Likert scales for patients to rate their music experience.

Music, when present, will be delivered via a speaker system allowing for communication between the urologist and the patient during the procedure. Only one urologist will be performing all flexible cystoscopies. Aside from the addition of music therapy for groups 1 and 2, standard of care will not be impacted.

Statistical analysis will be conducted by two-way ANCOVA comparing the mean of quantitative outcome variables between the three music groups and each sex. In the event of a significant interaction between the music and sex variables, one way-ANCOVA will be performed within each sex, followed by Bonferroni-corrected post-hoc tests.

All data will be collected and stored appropriately as according to institutional policies as well as any relevant chapters and sections of TCPS2.

Power analysis was performed to estimate the minimum sample size required to conduct the proposed ANCOVA analyses. A review of relevant literature indicated effect sizes ranging from small to large for both VAS and STAI scores. We therefore estimated our sample size using a medium effect size to provide a reasonable common ground among findings in the literature. Due to the 1:1:1 design for both sexes, we will target a sample size of 162 to allow for an equal allocation of 27 participants per group.

ELIGIBILITY:
Inclusion Criteria:

* All outpatient men and women needing diagnostic or surveillance flexible cystoscopy.
* 40 years or older.
* Presenting to outpatient urology clinic.

Exclusion Criteria:

* Narcotics/analgesics within the past 24 hours
* Stricture/anatomic urethra problems
* Current UTI
* Inability to complete survey or comply with experimental methods,
* Refusal to participate
* Rigid cystoscopy
* Manipulation during cystoscopy (stent removal, fulguration tumor, etc)
* Pre-existing chronic pelvic pain condition/diagnosis

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a 1:1:1 randomization with equal group membership performed for both male and female sexes - The envelopes will be randomized by pre-assigning an order of participants to each of the three groups within each sex using a Random sequence generator.
  This design is to appropriately account for potential differences in cystoscopy experience for males and females, due to differences in ureter length and anatomy.
Enrollment: 162 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Post-Cystoscopy Anxiety Score | Immediately after the procedure
  Anxiety score is measured using the State Trait Anxiety Inventory (STAI). The STAI consists of two questionnaires that classifies a patient's anxiety into three groups on a scale of 20 to 80. The STAI includes two component questionnaires known as State Anxiety and Trait Anxiety. Trait Anxiety corresponds with stable individual anxiety measures while State Anxiety refers to anxiety that an individual is experiencing at a specific given moment at time. As described by the State-Trait Anxiety Inventory for Adults manual, people with higher Trait Anxiety measures may have elevated State Anxiety measures as compared to people with lower Trait Anxiety. In our study, Trait Anxiety will be controlled for, since differences in Trait Anxiety may confound State Anxiety measurements due to the individual being naturally more anxious due to unrelated reasons. A higher STAI anxiety score indicates higher anxiety.
Change in Anxiety Score from immediately before to immediately after cystoscopy (delta STAI) | Change from immediately before the procedure to immediately after the procedure
  The delta State Trait Anxiety Inventory (delta STAI) is a measure of the change in STAI anxiety score immediately after the cystoscopy minus STAI anxiety score immediately prior to the cystoscopy. The delta STAI ranges on a scale from negative 60 to positive 60. A positive delta STAI score indicates that there was a greater STAI anxiety score immediately after the procedure as compared to immediately before the procedure. A higher positive delta STAI score means a greater increase in anxiety as compared to a lower delta STAI score. A negative delta STAI score indicates that there was a lower STAI anxiety score immediately after the procedure as compared to immediately before the procedure. A more negative delta STAI score indicates a greater decrease in anxiety as compared to a less negative delta STAI score. A delta STAI score of 0 indicates that there was no change in STAI anxiety score from immediately before the procedure to immediately after the procedure.
Pelvic pain score | Immediately after the procedure
  Pelvic pain will be measured using a Visual Analog Scale (VAS). The VAS score is completed by the patient ranking their pain intensity on 10-cm lines and providing a range of scores from 0 to 100. This measure is then converted to a score of 10 (to 1 decimal eg. 8.2/10). For this study, VAS scales will be filled out by the patient immediately following their cystoscopy. A higher VAS score indicates greater self reported pelvic pain.

SECONDARY OUTCOMES:
Pelvic discomfort score | Immediately after the procedure
  Pelvic discomfort will be measured using a Visual Analog Scale (VAS). The VAS score is completed by the patient ranking their discomfort on 10-cm lines and providing a range of scores from 0 to 100. This measure is then converted to a score of 10 (to 1 decimal eg. 8.2/10). For this study, VAS scales will be filled out in the post-procedure questionnaire by the patient immediately following their cystoscopy. A higher VAS score indicates greater self reported pelvic discomfort.
Patient satisfaction score | Immediately after the procedure
  Patient satisfaction with cystoscopy will be measured using a Visual Analog Scale (VAS). The VAS score is completed by the patient ranking their satisfaction on 10-cm lines and providing a range of scores from 0 to 100. This measure is then converted to a score of 10 (to 1 decimal eg. 8.2/10). For this study, VAS scales will be filled out in the post-procedure questionnaire by the patient immediately following their cystoscopy. A higher VAS score indicates greater self reported patient satisfaction.
Willingness to repeat cystoscopy score | Immediately after the procedure
  Willingness to repeat cystoscopy will be measured using a Visual Analog Scale (VAS). The VAS score is completed by the patient ranking their willingness to repeat cystoscopy on 10-cm lines and providing a range of scores from 0 to 100. This measure is then converted to a score of 10 (to 1 decimal eg. 8.2/10). For this study, VAS scales will be filled out in the post-procedure questionnaire by the patient immediately following their cystoscopy. A higher VAS score indicates greater willingness to repeat cystoscopy.
How pleasant patients from music intervention groups found the music | Immediately after the procedure
  How pleasant patients found the music during their cystoscopy will be measured using a 5-point Likert scale where patients rate their agreement with the statement "I found the music pleasant". Ratings include "Strongly agree, Agree, Neither agree nor disagree, Disagree, Strongly disagree".
How calming patients from music intervention groups found the music | Immediately after the procedure
  How calming patients found the music during their cystoscopy will be measured using a 5-point Likert scale where patients rate their agreement with the statement "I found the music calming". Ratings include "Strongly agree, Agree, Neither agree nor disagree, Disagree, Strongly disagree".
How much patients from music intervention groups found that music helped distract them from the cystoscopy procedure | Immediately after the procedure
  How distracting patients found the music during their cystoscopy will be measured using a 5-point Likert scale where patients rate their agreement with the statement "The music helped distract me from the cystoscopy procedure". Ratings include "Strongly agree, Agree, Neither agree nor disagree, Disagree, Strongly disagree".

CONTACTS AND LOCATIONS:
Overall Officials: Gavin M Langille, MD, Principal Investigator — Horizon Health Network, Dalhousie University Department of Urology
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No